CLINICAL TRIAL: NCT04182685
Title: Evaluation of Medical Conditions Associated With Zika Virus Infection in Managua, Nicaragua
Status: Completed | Type: Observational
Sponsor: RTI International (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of North Carolina, Chapel Hill (Other); Sustainable Sciences Institute (Managua, Nicaragua) (Unknown); Ministry of Health Nicaragua (Unknown)
Responsible Party: Sponsor
Other Study IDs: CNDR CIRE-16/07/19-099.Ver2; 1R21HD095420-01A1 (NIH)
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Zika Virus
Keywords: Zika virus; neurodevelopment; neurological sequelae
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ZIKV-exposed children: Children age 5-15 with a positive Zika virus PCR test result.
- ZIKV-unexposed children: Children age 5-15 who have not had a Zika virus infection as determined by serological assays.

SUMMARY:
Zika virus (ZIKV) infection spread throughout the Americas with devastating consequences. Recent limited evidence suggests the potential for neurological effects associated with postnatally acquired ZIKV infection in humans; however, the impact on children is unknown. The researchers will conduct a longitudinal study of approximately 450 Nicaraguan children who were ages 2-12 in 2016 to evaluate the presence and persistence of neurological symptoms associated with ZIKV infection and to test whether ZIKV-infected children are at greater risk for developing neurological outcomes compared to uninfected children.

DETAILED DESCRIPTION:
In 2016, the World Health Organization designated the Zika virus (ZIKV) epidemic as a Public Health Emergency of International Concern because of the emerging association between microcephaly and ZIKV infection during pregnancy. Although many studies have evaluated the biochemical pathways for congenital ZIKV infection and related severe neurodevelopmental fetal and neonatal outcomes, research on health outcomes related to postnatally acquired ZIKV infection in children is lacking. The few existing epidemiological reports describe incidence rates of acquired ZIKV infection among symptomatic children only, and they predominantly include probable cases based on clinical signs and symptoms. Case reports and surveillance of acute central nervous system disease in adults and adolescents secondary to ZIKV infection suggest that ZIKV may have a broader impact on neurological health beyond that observed in congenitally exposed newborns, including neuropsychological deficits, long-term fatigue, and spinal cord lesions with unilateral paresthesia and muscle weakness. The neurotropic properties of ZIKV and its impact on developing neural cells in postnatally infected mice and nonhuman primates also raise concerns about the potential neurological sequelae of postnatal ZIKV infection, particularly in children. However, the extent to which acquired ZIKV infection can negatively affect the nervous systems and cause long-term neurological damage or cognitive effects is currently unknown. Although the existing evidence is limited, it provides the scientific premise for the hypothesis that ZIKV-infected children are at greater risk for developing neurological sequelae (e.g., cognitive, behavioral, sensory, motor deficits) compared to uninfected children. The researchers will conduct a longitudinal study of approximately 450 Nicaraguan children in the Pediatric Dengue Cohort Study (PDCS) who were ages 2- 12 during January 2016-January 2017, with and without acquired ZIKV infection, to accomplish the following aims:

Aim 1: Evaluate the presence and persistence of neurological symptoms among children with acquired ZIKV infection. Children from the PDCS who presented to a local clinic with ZIKV-like symptoms from January 2016 through January 2017 were tested for ZIKV and given a baseline symptoms questionnaire that included neurological symptoms (e.g., seizures, headaches, muscle weakness, fatigue). The researchers will enroll 225 symptomatic ZIKV-infected children who were ages 2-12 during that time period and give them the same symptoms questionnaire at a follow-up visit in 2019. The researchers will analyze the baseline and follow-up symptoms data to evaluate ZIKV-associated neurological symptom severity and persistence.

Aim 2: Test for associations between neurological sequelae and acquired ZIKV infection.

Hypothesis: ZIKV-infected children are at greater risk for developing neurological sequelae (e.g., cognitive, behavioral, sensory, and motor deficits) compared to uninfected children. The researchers will enroll an equal number of ZIKV-uninfected PDCS children matched by age and sex to the ZIKV-infected children described in Aim 1 to provide a comparison group. For both ZIKV-infected and uninfected children, at the 2019/2020 study visit, the researchers will assess (1) clinical indicators of neurological impairment (e.g., vision, hearing, motor, and sensory functioning) by direct observation; (2) functioning across a wide range of domains (e.g., executive function, visual-spatial thinking, processing speed, attention, adaptive behavior) by administering a comprehensive neuropsychological assessment battery; and (3) factors related to neurological functioning (e.g., mood and sleep disorders).

The researchers will use regression models to calculate relative risks and 95% confidence intervals for the relationship between ZIKV status, clinical indicators of neurological impairment, and neuropsychological functioning across a wide range of domains. Additionally, we the researchers will assess the role of sex as a biological variable in stratified analyses. By leveraging the existing PDCS cohort and locally tested neurodevelopmental assessment tools, our cost-effective the study will provide invaluable information for determining the merit of conducting a larger and more in-depth study of the neurological impacts of acquired ZIKV infection that could be used to inform clinical practice and support the establishment of school-based educational interventions for affected children.

ELIGIBILITY:
Inclusion Criteria:

* 5-15 years of age at the time of enrollment;
* Active in the PDCS
* Complete data on age, sex, and ZIKV status;
* Willingness to participate in the study visit;
* Written parental permission and assent to participate, as appropriate by age.

Exclusion Criteria:

* Children with evidence in their medical charts of a diagnosis of a neurological (e.g., traumatic brain injuries, seizure disorder, stroke) or neurodevelopmental disorder (e.g., ADHD, Autism, Intellectual Disability) before January 2016.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study participants will be recruited from the Pediatric Dengue Cohort Study (PDCS). The PDCS is based out of the HCSFV, the primary public health center for District II of Managua serving a catchment area of more than 60,000 people. Currently, there are 3,818 active participants in the cohort. PDCS children who presented to HCSFV with fever or illness between January 2016 and January 2017 were tested for ZIKV by RT-PCR. The RT-PCR test results define ZIKV exposure in this study. All children in the cohort come to HCSFV once a year to provide a blood sample, regardless of symptoms.
  In 2016 and 2017, these specimens were tested for ZIKV infection using a nonstructural protein 1 (NS1) blockade-of-binding (BOB) ELISA assay for ZIKV. The results of this serological assay define the ZIKV-unexposed population in this study. See 'Eligibility Criteria' for additional information.
Sampling Method: Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of short-term self-reported neurological symptoms among ZIKV-exposed | Baseline data were collected at the time of infection between January 2016 and January 2017
  When ill children presented to the Health Center Socrates Flores Vivas (HCSFV) between January 2016 and January 2017, they were tested for Zika virus at that visit and 14-21 days later. A questionnaire was administered to the parent/guardian of the child at both the initial and convalescent visits to ascertain information about the child's recent neurological symptoms (i.e., persistent headaches, muscle weakness, seizures, fainting/blackouts, lethargy/fatigue, and back pain). Self-reported outcome.
Prevalence of short-term clinically-observed neurological symptoms among ZIKV-exposed | Baseline data were collected at the time of infection between January 2016 and January 2017
  When ill children presented to the Health Center Socrates Flores Vivas (HCSFV) between January 2016 and January 2017, they were tested for Zika virus at that visit and 14-21 days later. An extensive clinical exam was conducted at both the initial and convalescent visits to assess neurological symptoms (i.e., paralysis, paresthesia, limb weakness).
Incidence of long-term clinically-observed neurological sequelae | Current study visit (between October 2019-December 2020)
  At the current study visit, for both ZIKV-infected and uninfected children, a pediatrician will conduct a neurological exam to assess cranial nerve function and to look for evidence of neurological impairment (e.g., vision, hearing, motor, and sensory impairment).
Incidence of long-term self-reported neurological sequelae | Current study visit (between October 2019-December 2020)
  A neurological symptoms questionnaire will be administered by a pediatrician during the clinical exam to ascertain information about neurological symptoms (i.e., paralysis, paresthesia, persistent headaches, muscle weakness, seizures, fainting/blackouts, lethargy/fatigue, and back pain) in the last 6 months. The questionnaire also collects information about changes in vision, hearing, and motor function, as well as difficulty concentrating and fatigue, since January 2016. Patient-reported outcome.
Neurocognitive function | Current study visit (between October 2019-December 2020)
  Bateria IV Woodcock-Munoz Cognitive module will be administered by a psychologist to assess neurocognitive functioning. The Bateria IV Woodcock-Munoz assesses comprehension-knowledge, visual-spatial thinking, auditory processing, processing speed, memory, attention, and fluid reasoning. Test scores less than one standard deviation from the instrument's normed mean will be considered 'at-risk' for neurocognitive deficiencies.
Nonverbal Intelligence | Current study visit (between October 2019-December 2020)
  The Test of Nonverbal Intelligence 4, which assesses intelligence, aptitude, abstract reasoning, and problem solving with minimal physical response, will be administered by a psychologist. Test scores less than one standard deviation from the instrument's normed mean will be considered 'at-risk' for cognitive deficiency.
Behavioral problems | Current study visit (between October 2019-December 2020)
  The Child Behavior Checklist (CBCL) will be administered to the parent/guardian of the child participant to ascertain information about the child's behavior. The CBCL provides a score of Internalizing, Externalizing, and Total Behavior Problems, along with eight clinical domains. Children with scores less than two standard deviations from the test normed mean will be considered 'at-risk' for behavioral problems.

SECONDARY OUTCOMES:
Depression | Current study visit (between October 2019-December 2020)
  The Children's Depression Inventory Short Form will be administered to the child by a psychologist to obtain information about depression in children age 7-15. Scores range from 0 to 20 with higher scores indicating more severe depression symptoms. Self-reported outcome.
Anxiety | Current study visit (between October 2019-December 2020)
  The Spence Children's Anxiety Scales will be administered to the child by a psychologist to obtain information about anxiety in children age 7-15. The scale assesses six domains of anxiety including generalized anxiety (score rang 0-18), panic/agoraphobia (score range 0-27), social phobia (score range 0-18), separation anxiety (score range 0-18), obsessive compulsive disorder (score range 0-18), and physical injury fears (score rang 0-15). Higher scores indicate more severe anxiety. Self-reported outcome.
Sleep problems | Current study visit (between October 2019-December 2020)
  The BEARS sleep questionnaire will be administered to the child, if age 13 or older, or the parent/guardian, if the child is age 12 or younger, to obtain information about disordered sleeping. Self-reported outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jill F. Lebov, PhD, Principal Investigator — RTI International
Locations (1):
- Health Center Socrates Flores Vivas, Managua, Nicaragua

REFERENCES:
- [Background] Schrank FA, McGrew KS, Ruef ML, Alvarado CG. Batería III Woodcock-Muñoz™. Assessment Service Bulletin. 2005(1).
- [Background] Achenbach TM, Ruffle TM. The Child Behavior Checklist and related forms for assessing behavioral/emotional problems and competencies. Pediatr Rev. 2000 Aug;21(8):265-71. doi: 10.1542/pir.21-8-265. No abstract available. PMID 10922023
- [Background] Brown L, Sherbenou RJ, Johnsen SK. TONI-4, Test of Nonverbal Intelligence. Pro-ed; 2010.
- [Background] Davanzo P, Kerwin L, Nikore V, Esparza C, Forness S, Murrelle L. Spanish translation and reliability testing of the Child Depression Inventory. Child Psychiatry Hum Dev. 2004 Fall;35(1):75-92. doi: 10.1023/b:chud.0000039321.56041.cd. PMID 15626326
- [Background] Orgiles M, Mendez X, Spence SH, Huedo-Medina TB, Espada JP. Spanish validation of the Spence Children's Anxiety Scale. Child Psychiatry Hum Dev. 2012 Apr;43(2):271-81. doi: 10.1007/s10578-011-0265-y. PMID 22086155
- [Background] Mindell, J.A, and Owens, J. O. A Clinical Guide to Pediatric Sleep: Diagnosis and Management of Sleep Problems. Lippincott Williams & Wilkins, 2015.